CLINICAL TRIAL: NCT01450397
Title: MRI Results in Dupuytren's Contracture Before and After Injection With Xiaflex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Auxilium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11052
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Dupuytren's Disease
Keywords: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase; Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XIAFLEX (Other): XIAFlEX
  Interventions: Biological: XIAFLEX

INTERVENTIONS:
Biological: XIAFLEX — One Injection of 0.58 mg of Xiaflex into the affected area of the hand.
  Other Names: Collagenase

SUMMARY:
The purpose of this study is to determine the effects of XIAFLEX on your finger through MRI.

DETAILED DESCRIPTION:
Collagenase injections for the treatment of Dupuytren's Contracture is a newly approved protocol which has shown early efficacy. There are very few studies which examine the MRI appearance of Dupuytren's disease. There are no studies that evaluate the condition of the cord after collagenase injection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Dupuytren's Disease affecting only the metacarpophalangeal joint of the 4th or 5th finger.
* Subject has only one finger affected by the disease.
* Patients will be 35 years of age of older.
* Patients will be able to read, speak, and understand English or have available adequate translation assistance and be able to provide voluntary written consent to participate.

Exclusion Criteria:

* Female patients who are nursing or pregnant, or plan to become pregnant during the treatment phase.
* Patient has a chronic muscular, neurological or neuromuscular disorder that affects the hands.
* Patient has known allergy to collagenase or any other excipient of Xiaflex.
* Patient has received any collagenase treatments before the first dose of Xiaflex.
* Patient with abnormal coagulation, including patients who have received anticoagulant medications other than low-dose aspirin within 7 days of the injection.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Wolfe, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hosptial for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from July 2011 to December 2011. Enrollment was completed in a medical clinic.
Groups:
- XIAFLEX: 0.58 mg of Xiaflex injected into a palpable Dupuytren's cord
Period: Overall Study
Arm/Group | XIAFLEX
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- XIAFLEX: Patient who have received XIAFLEX
Arm/Group | XIAFLEX
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: The Measured Change in Volume of the Cord by MRI Before and After XIAFLEX Injection and Manual Manipulation.
Description: Change in Volume (millimeter cubed) of the Cord by MRI between Baseline and 30 days after XIAFLEX injection and manual manipulation.
Time Frame: Baseline and 30 days
Measure: Mean (Full Range); unit: mm^3
Groups:
- XIAFLEX: Subjects receiving one Xiaflex injection
Arm/Group | XIAFLEX
Number analyzed (Participants) | 5
mm^3 | 482 [188 to 670]
Statistical Analysis 1: Comparison: XIAFLEX; Test type: Superiority or Other; p < 0.0013, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- XIAFLEX: Patient who received XIAFLEX
Arm/Group | XIAFLEX
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No